CLINICAL TRIAL: NCT04617535
Title: Compassionate Use of REGN-COV2 for the Treatment of COVID-19
Status: No longer available | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R10933-10987-COV
Record Dates: First submitted 2020-11-02; First posted 2020-11-05 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
Keywords: Post-exposure
MeSH Terms: conditions — COVID-19 | interventions — casirivimab and imdevimab drug combination; casirivimab; imdevimab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: REGN10933+REGN10987 combination therapy — Administered intravenously (IV) single dose
  Other Names: REGN-COV2; Casirivimab; Imdevimab; REGEN-COV™; Ronapreve™

SUMMARY:
Compassionate Use requests will be considered for individuals who test positive for SARS-CoV-2 and where there is reasonable basis to believe that the patient is infected with a susceptible variant.

DETAILED DESCRIPTION:
Compassionate Use requests are only being considered in response to Individual Patient Investigational New Drug (IND) applications.

Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343